CLINICAL TRIAL: NCT06000592
Title: Safety, Feasibility, and Efficacy of Transcutaneous Spinal Cord Stimulation on Stabilizing Blood Pressure for Acute Inpatients With Spinal Cord Injury
Brief Title: Safety, Feasibility, and Efficacy of TSCS on Stabilizing Blood Pressure for Acute Inpatients With SCI
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Jill M. Wecht, Ed.D. (U.S. Federal Agency)
Collaborators: Icahn School of Medicine at Mount Sinai (Other)
Responsible Party: Sponsor-Investigator, Jill M. Wecht, Ed.D., Research Health Scientist, James J. Peters Veterans Affairs Medical Center
Organization: James J. Peters Veterans Affairs Medical Center (U.S. Federal Agency)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 1648740
Record Dates: First submitted 2023-06-23; First posted 2023-08-21 (Actual); Last update posted 2024-04-02 (Actual); Status verified 2024-04

CONDITIONS: Acute Spinal Cord Injury; Spinal Cord Injuries; Neuromodulation; Traumatic Spinal Cord Injury; Spinal Cord Stimulation; SCI - Spinal Cord Injury; Blood Pressure; Blood Pressure Disorders
MeSH Terms: conditions — Spinal Cord Injuries

STUDY DESIGN:
Masking Description: Participant awareness during TSCS appears to be unavoidable. The FDA recognizes that some trials of non-pharmacological interventions cannot be fully shammed or blinded, yet with careful blinding of data assessors, it is possible to obtain reliable results that meet FDA approval criteria.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (1):
- transcutaneous spinal stimulation (Experimental): Transcutaneous spinal cord stimulation (TSCS) protocol to stabilize seated systolic blood pressure in newly injured patients with spinal cord injury and to test the ability of TSCS to reduce the fall in blood pressure when these patients are moved from the supine to the seated position.
  Interventions: Device: Digitimer

INTERVENTIONS:
Device: Digitimer — transcutaneous spinal cord stimulation for blood pressure control following spinal cord injury.

SUMMARY:
Current forms of pharmacologic and non-pharmacologic treatments for hypotension and orthostatic hypotension (OH) remain inadequate during acute inpatient rehabilitation (AIR) following a traumatic spinal cord injury (SCI). A critical need exists for the identification of safe, practical, and effective treatment options that stabilize blood pressure (BP) after traumatic SCI. Recent published evidence suggests that transcutaneous Spinal Cord Stimulation (TSCS) can be used to raise seated BP, and mitigate the falls in BP during orthostatic repositioning in individuals with chronic SCI. This site-specific project will focus on the use of TSCS to stabilizing seated BP and mitigate the fall in BP during orthostatic repositioning during AIR following traumatic SCI.

DETAILED DESCRIPTION:
Based on available evidence, TSCS may have advantages over current pharmacological approaches to the treatment of hypotension and OH: (1) does not exacerbate polypharmacy, (2) can be activated/deactivated rapidly, and (3) can be applied in synergy with physical exercise. TSCS represents an alternate approach to epidural SCS, with far greater potential to reach large numbers of individuals, thus providing for a greater likelihood of clinical implementation with fewer risk. We are asking several key questions: (1) what are the effects of TSCS on seated BP and BP changes during an orthostatic challenge, (2) is the application of TSCS during AIR tolerable based on pain reporting, (3) is there evidence of superficial burns to the skin near the site of cathode or anode placement, and (4) are the symptoms of orthostatic intolerance reduced with TSCS? To facilitate adoption of TSCS for widespread clinical use, we have designed a spatial-temporal mapping and parameter configuration approach that will result in a key deliverable for SCI care: a standard, easy to follow algorithm that will maximize individual benefits of spinal neuromodulation, while minimizing the burden on healthcare professionals. This project will provide the foundational evidence to support the feasible and safe application of TSCS for widespread clinical utility in the newly injured SCI population, thereby overcoming barriers to engagement in prescribed AIR regimens that are imposed by autonomic nervous system dysfunction.

ELIGIBILITY:
Inclusion Criteria:

* Newly injured patients with traumatic SCI
* Admitted to Acute Inpatient Rehabilitation at Mount Sinai
* Within one year of SCI
* Seated hypotension (systolic BP ≤ 110 mmHg for males or ≤ 100 mmHg for females)
* Orthostatic hypotension (fall in systolic BP ≥ 20 mmHg and/or a fall in diastolic BP ≥ 10 mmHg within 10 minutes of assuming an upright position)
* Daily fluctuation in systolic BP ≥ 20 mmHg and/or fluctuation in diastolic BP ≥ 10 mmHg
* At least 14 years old

Exclusion Criteria:

* Implanted brain/spine/nerve stimulators
* Cochlear implants
* Cardiac pacemaker/defibrillator, or intracardiac lines
* Open skin lesions on or near the electrode placement sites (neck, upper back)
* Significant coronary artery or cardiac conduction disease
* Recent history of myocardial infarction
* Insufficient mental capacity to understand and independently provide consent
* Pregnancy
* Cancer
* Deemed unsuitable by study physician

Ages: 14 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2022-01-01 (Actual); Primary Completion 2026-08-31 (Estimated); Study Completion 2026-10-01 (Estimated)

PRIMARY OUTCOMES:
The efficacy (#1) of TSCS to improve autonomic control following acute SCI. | Acute Inpatient Rehabilitation following SCI (up to 4 months)
  Blood pressure changes (mmHg) during the sit-up test with TSCS compared to no stimulation.
The safety (#1) of TSCS to improve autonomic control following acute SCI. | Acute Inpatient Rehabilitation following SCI (up to 4 months)
  Assess pain levels using a Likert Scale 0-10 (0=no pain, 10=worst pain).
The safety (#2) of TSCS to improve autonomic control following acute SCI. | Acute Inpatient Rehabilitation following SCI (up to 4 months)
  Document any skin changes (burns) following use of TSCS in count of occurrences.

SECONDARY OUTCOMES:
The efficacy (#2) of TSCS to improve autonomic control following acute SCI. | Acute Inpatient Rehabilitation following SCI (up to 4 months)
  To compare dizziness symptoms on a Likert Scale 0-10 (0=no dizziness, 10=worst dizziness) during the sit-up test with TSCS compared to no stimulation..

CONTACTS AND LOCATIONS:
Overall Officials: Thomas N Bryce, MD, Study Director — Icahn School of Medicine at Mount Sinai
Locations (1):
- The Icahn School of Medicine at Mount Sinai, New York, New York, United States